CLINICAL TRIAL: NCT00372060
Title: MK0431 (Sitagliptin) Phase III Clinical Study -Pioglitazone add-on Study for Patients With Type 2 Diabetes Mellitus
Brief Title: MK0431 (Sitagliptin) Pioglitazone Add-on Study for Patients With Type 2 Diabetes Mellitus (0431-055)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-055; 2006_029
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK0431 + pioglitazone
  Interventions: Drug: sitagliptin phosphate; Drug: Comparator: pioglitazone
- 2 (Placebo Comparator): Placebo/MK0431 + pioglitazone
  Interventions: Drug: Comparator: sitagliptin phosphate (MK0431); Drug: Comparator: pioglitazone; Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: sitagliptin phosphate — Sitagliptin (MK0431) 50 or 100 mg once daily for 52 weeks
  Other Names: MK0431
  Arms: 1
Drug: Comparator: sitagliptin phosphate (MK0431) — Sitagliptin (MK0431) 50 or 100 mg once daily for 40 weeks
  Other Names: MK0431
  Arms: 2
Drug: Comparator: pioglitazone — pioglitazone once daily for 52 weeks
Drug: Comparator: placebo (unspecified) — Placebo once daily for 12 weeks
  Arms: 2

SUMMARY:
The clinical study determines the safety and efficacy of MK0431 in patients with type 2 diabetes mellitus who have inadequate glycemic control on pioglitazone as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients Have Type 2 Diabetes Mellitus
* On Diet/Exercise Therapy And Pioglitazone As Monotherapy

Exclusion Criteria:

* Patients Have Type 1 Diabetes Mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2006-08-21 (Actual); Primary Completion 2008-02-05 (Actual); Study Completion 2008-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Kashiwagi A, Kadowaki T, Tajima N, Nonaka K, Taniguchi T, Nishii M, Ferreira JC, Amatruda JM. Sitagliptin added to treatment with ongoing pioglitazone for up to 52 weeks improves glycemic control in Japanese patients with type 2 diabetes. J Diabetes Investig. 2011 Oct 7;2(5):381-90. doi: 10.1111/j.2040-1124.2011.00120.x. PMID 24843518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III.
  Date of first patient in: 22 August 2006. Date of last patient's last visit for Period I: 1 May 2007.
  Date of last patient's last visit for Period II: 5 February 2008. Number of randomized patients: 134.
  The study was conducted at 32 centers in Japan.
Pre-assignment Details: Following a screening period of at least 4 weeks and a 2 or 8-week observation period, patients who were on pioglitazone monotherapy for at least 8 weeks and met all other entry criteria were randomized to receive: sitagliptin/sitagliptin or placebo/sitagliptin.
  The starting dose of sitagliptin was 50 mg for all patients.
Groups:
- Sitagliptin / Sitagliptin: The Sitagliptin/Sitagliptin group includes data from all patients randomized to receive treatment with sitagliptin (Weeks 0-52) and pioglitazone (Weeks 0-52) orally once daily. Includes patients who received only sitagliptin 50 mg and those who started on sitagliptin 50 mg and whose dose was subsequently up-titrated to sitagliptin 100 mg orally once daily. Uptitration of sitagliptin dose was to occur for patients with FPG >140 mg/dL at any time from Week 16 to Week 40 or HbA1c values >7.0% at any time from Week 24 to Week 40. The sitagliptin dose was to have remained stable after Week 40.
- Placebo / Sitagliptin: The Placebo/Sitagliptin group includes data from all patients randomized to receive the sequence of placebo (Weeks 0-12) / sitagliptin (Weeks 12-52) and pioglitazone (Weeks 0-52) orally once daily. Includes patients who received only sitagliptin 50 mg and those who started on sitagliptin 50 mg and whose dose was subsequently up-titrated to sitagliptin 100 mg orally once daily. Uptitration of sitagliptin dose was to occur for patients with FPG >140 mg/dL at any time from Week 16 to Week 40 or HbA1c values >7.0% at any time from Week 24 to Week 40. The sitagliptin dose was to have remained stable after Week 40.
Period: Period I - Double-blind (Weeks 0-12)
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin
Started | 66 (The planned number of enrolled patients was 130. The actual number of enrolled patients was 134.) | 68
Completed | 63 | 67
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — No improvement in hyperglycemia | 1 | 0
Period: Period II - Open-label (Weeks 12-52)
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin
Started | 63 | 67
Completed | 49 | 59
Not Completed | 14 | 8
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 9 | 8
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.9) | 59.0 (9.2) | 58.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 47
  Male | 38 | 49 | 87
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 146.8 (33.1) | 151.3 (34.6) | 149.1 (33.8)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.7 (0.9) | 7.6 (0.8) | 7.7 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c ) at Week 12
Description: Change from the baseline measurement, where the baseline measurement was obtained at randomization (0 week) before receiving study medication.
Time Frame: 12 Weeks
Population: Analysis in the Full Analysis Set with Last Observation Carried Forward (The Full Analysis Set population includes all randomized patients who took at least 1 dose of study medication and had both a baseline and at least one post-baseline value.)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin
Number analyzed (Participants) | 66 | 68
Percent | -0.4 [-0.6 to -0.3] | 0.4 [0.3 to 0.5]
Statistical Analysis 1: Comparison: Sitagliptin / Sitagliptin vs Placebo / Sitagliptin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior oral anti-hyperglycemic medication (except for pioglitazone), and baseline HbA1c; Least-squares Mean Difference = -0.8, 95% CI [-1.0 to -0.6], Standard Error of Mean 0.10

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: Change from baseline measurement, where the baseline measurement was obtained at randomization (0 week) before receiving study medication.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin
Number analyzed (Participants) | 66 | 68
mg/dL | -12.2 [-17.0 to -7.5] | 4.4 [-0.3 to 9.1]
Statistical Analysis 1: Comparison: Sitagliptin / Sitagliptin vs Placebo / Sitagliptin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior oral anti-hyperglycemic medication (except for pioglitazone), and baseline fasting plasma glucose; Least-squares Mean Difference = -16.7, 95% CI [-23.4 to -10.0], Standard Error of Mean 3.39

3. Other Pre Specified Outcome: Change From Baseline in 2 Hour Postprandial Glucose at Week 12
Description: as for outcome 2
Time Frame: 12 weeks
Population: Analysis in the Full Analysis Set without Last Observation Carried Forward (The Full Analysis Set population includes all randomized patients who took at least 1 dose of study medication and had both a baseline and at least one post-baseline values.).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin
Number analyzed (Participants) | 63 | 67
mg/dL | -42.7 [-53.7 to -31.7] | 6.4 [-4.2 to 17.1]
Statistical Analysis 1: Comparison: Sitagliptin / Sitagliptin vs Placebo / Sitagliptin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior oral anti-hyperglycemic medication (except for pioglitazone), and baseline 2-hour postprandial glucose; Least-squares Mean Difference = -49.2, 95% CI [-64.5 to -33.9], Standard Error of Mean 7.7

4. Other Pre Specified Outcome: Change From Baseline in Hemoglobin A1c (HbA1c ) at Week 52
Description: Change from the last value before receiving sitagliptin therapy: Week 0 for Sitagliptin/Sitagliptin group and Week 12 for the Placebo/Sitagliptin group.
Time Frame: Week 52 (reflecting change from Week 0) for Sitagliptin/Sitagliptin group; Weeks 52 (reflecting change from Week 12) for Placebo/Sitagliptin group.
Population: The Completers Population (CP) includes all randomized patients who took at least 1 dose of sitagliptin and had [1] a baseline (Sitagliptin/Sitagliptin group) or Week 12 (Placebo/Sitagliptin group) value and [2] a value at Week 52.
Measure: Mean (95% Confidence Interval); unit: Percent
Groups:
- Sitagliptin / Sitagliptin: The Sitagliptin/Sitagliptin group includes data from all patients randomized to receive treatment with sitagliptin (Weeks 0-52) orally once daily who were in the CP. This column of data reflects the change from Week 0 at Week 52.
- Placebo / Sitagliptin: The Placebo/Sitagliptin group includes data from all patients randomized to receive the sequence of placebo (Weeks 0-12) / sitagliptin (Weeks 12-52) orally once daily and who received at least one dose of sitagliptin and were in the CP. This column of data reflects the change from Week 12 at Week 52.
Arm/Group | Sitagliptin / Sitagliptin | Placebo / Sitagliptin
Number analyzed (Participants) | 50 | 59
Percent | -0.6 [-0.8 to -0.5] | -0.9 [-1.1 to -0.7]

ADVERSE EVENTS:
Groups:
- Sitagliptin/Sitagliptin (Data Through Week 12): The Sitagliptin/Sitagliptin group includes data from all patients randomized to receive treatment with sitagliptin orally once daily (Weeks 0-52). This column of data includes only Weeks 0-12.
- Placebo/Sitagliptin (Data Through Week 12): The Placebo/Sitagliptin group includes data from all patients randomized to receive the sequence of placebo (Weeks 0-12) / sitagliptin (Weeks 12-52) orally once daily. This column of data includes only Weeks 0-12.
- Pooled Sitagliptin (Data Through Week 52): The Pooled Sitagliptin group includes data from all patients who took sitagliptin in either treatment group. Includes data from Week 0 to Week 52 for patients in the Sitagliptin/Sitagliptin group and data from Week 12 to Week 52 for patients in the Placebo/Sitagliptin group. Includes patients (from either group) who received only sitagliptin 50 mg and those who started on sitagliptin 50 mg and whose dose was subsequently up-titrated to sitagliptin 100 mg orally once daily.
Arm/Group | Sitagliptin/Sitagliptin (Data Through Week 12) | Placebo/Sitagliptin (Data Through Week 12) | Pooled Sitagliptin (Data Through Week 52)
Serious Adverse Events (participants affected / at risk) | 3 | 1 | 7
Other Adverse Events (participants affected / at risk) | 21 | 23 | 80
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin/Sitagliptin (Data Through Week 12) | Placebo/Sitagliptin (Data Through Week 12) | Pooled Sitagliptin (Data Through Week 52)
Coronary artery stenosis (Cardiac disorders) | 1/66 | 0/68 | 1/133
Enteritis infectious (Infections and infestations) | 0/66 | 0/68 | 1/133
Patella fracture (Injury, poisoning and procedural complications) | 0/66 | 0/68 | 1/133
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0/66 | 0/68 | 1/133
Rib fracture (Injury, poisoning and procedural complications) | 0/66 | 0/68 | 1/133
Ligament injury (Injury, poisoning and procedural complications) | 0/66 | 1/68 | 0/133
Lower limb fracture (Injury, poisoning and procedural complications) | 0/66 | 1/68 | 0/133
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/66 | 0/68 | 1/133
Cerebral infarction (Nervous system disorders) | 1/66 | 0/68 | 1/133
Hypertension (Vascular disorders) | 1/66 | 0/68 | 1/133
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin/Sitagliptin (Data Through Week 12) | Placebo/Sitagliptin (Data Through Week 12) | Pooled Sitagliptin (Data Through Week 52)
Periodontitis (Gastrointestinal disorders) | 0/66 | 0/68 | 7/133
Nasopharyngitis (Infections and infestations) | 11/66 | 17/68 | 48/133
Weight increased (Investigations) | 2/66 | 0/68 | 10/133
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/66 | 0/68 | 8/133
Hypoaesthesia (Nervous system disorders) | 0/66 | 2/68 | 7/133
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9/66 | 3/68 | 19/133
Blood creatine phosphokinase increased (Investigations) | 1/66 | 2/68 | 17/133

LIMITATIONS AND CAVEATS:
Period II (Weeks 12-52) was open-label and uncontrolled, with all patients receiving sitagliptin. Results are pooled data from both treatment groups and should be considered in the context of the Type 2 Diabetes Mellitus (T2DM) population studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.